CLINICAL TRIAL: NCT02870673
Title: Assessment of the Effectiveness of Ultrasound-guided Acupuncture in the Management of Carpal Tunnel Syndrome
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Taipei Medical University Hospital (Other)
Responsible Party: Principal Investigator, You-Jen Tang, Principal Investigator, Taipei Medical University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: N201605074
Record Dates: First submitted 2016-08-08; First posted 2016-08-17 (Estimated); Last update posted 2016-08-19 (Estimated); Status verified 2016-08

CONDITIONS: Carpal Tunnel Syndrome
Keywords: acupuncture; electrical stimulation; carpal tunnel syndrome
MeSH Terms: conditions — Carpal Tunnel Syndrome | interventions — Triamcinolone Acetonide; Lidocaine; Electroacupuncture

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Injection of Shincort 0.5 ml and Xylocaine 0.5ml mixture (Active Comparator): In the first week of recruitment, this group will receive the local injection around the distal wrist crease with mixture of Shincort Inj(10mg/ml) 0.5 ml and xylocaine(20mg/ml) 0.5 ml only one time.
  The ultrasound-guided procedure is performed by the orthopedic physician.
  Interventions: Drug: SHINCORT; Drug: XYLOCAINE
- sham electroacupuncture (Experimental): In this group, the participants receive acupuncture treatment and only 2 minutes electrical stimulation.
  Each needle insertion depth and position are confirmed by the ultrasound. The procedure makes sure that needle pin is directly placed on the median nerve and prevent nerve penetration. Then the electrical stimulator is connected to the needles as cathode and anode and is turned on to the intensity which can induce thenar muscle contraction or reach the upper limit of the participant. After 2 minutes, the stimulator will turn off spontaneously and the participant will not be informed.
  The whole course will cost 20 minutes after needles are pulled out. Every participant is asked to receive 1 treatment per week in the consecutive 3 months(total 12 times).
  Interventions: Device: sham electroacupuncture
- electroacupuncture (Experimental): In this group, the participants receive acupuncture treatment and 20 minutes electrical stimulation.
  Each needle insertion depth and position are confirmed by the ultrasound. The procedure makes sure that needle pin is directly placed on the median nerve and prevent nerve penetration. Then the electrical stimulator is connected to the needles as cathode and anode and is turned on to the intensity which can induce thenar muscle contraction or reach the upper limit of the participant.
  The whole course will cost 20 minutes after needles are pulled out. Every participant is asked to receive 1 treatment per week in the consecutive 3 months(total 12 times).
  Interventions: Device: electroacupuncture

INTERVENTIONS:
Drug: SHINCORT — triamcinolone Acetonide (10mg/ml) 0.5 ml
  Other Names: triamcinolone Acetonide
  Arms: Injection of Shincort 0.5 ml and Xylocaine 0.5ml mixture
Drug: XYLOCAINE — xylocaine(20mg/ml) 0.5 ml
  Other Names: XYLOCAINE IV INJECTION
  Arms: Injection of Shincort 0.5 ml and Xylocaine 0.5ml mixture
Device: sham electroacupuncture — 1.5 inches 32 gauze stainless steel needles Transcutaneous electrical nerve stimulation machine (MODEL-05B(6))
  Arms: sham electroacupuncture
Device: electroacupuncture — 1.5 inches 32 gauze stainless steel needles Transcutaneous electrical nerve stimulation machine (MODEL-05B(6))
  Arms: electroacupuncture

SUMMARY:
In clinical practice, carpal tunnel syndrome (CTS) is the common disease of peripheral neuropathy and usually happened to female, mid-age population, overweight persons, and those who overused their hands for work or production. Some research claimed this might be correlated to anatomical characteristics such as the longer anteroposterior diameter or smaller cross section area of the wrist. Preliminary symptoms often start with sensory domain (pain, tingling, paresthesia and especially night awakening due to symptoms mentioned above) and then progress to motor domain (thenar muscle atrophy and clumsiness) if left untreated.

Depending on the severity, patient's willingness and convenience, there are many options for CTS. For those whose symptoms are mild to moderate, conservative therapies are usually the first choice, including physiotherapies, local injection and night splints. Local steroid is proven to be effective to relieve the symptoms of CTS shortly up to 3 months. However, the effects will decline gradually and repetitive injections is suggestive. The patients with severe symptoms which comprise thenar muscle atrophy will be advised to receive decompression surgery.the surgery can alleviate the illness with high success rate up to 70%. Unfortunately, there are still patients who will relapse or undergo side effects, for example, finger weakness.

In recent years, acupuncture researches focused on CTS intervention have been outgrowing and promising. Whereas, there are still lack of evidence which stands for the therapeutic effects comparing with local steroid injection. This limits the built-up of suspect mechanism of acupuncture intervention for CTS.

This is a preliminary, randomized and single-blinded study which started since 2016 and last for a year. The investigators utilize ultrasound to guide the depth of needle penetration which prevents unnecessarily tissues injury such as artery or dry needle injury. This procedure also guarantees the needles lie directly on the upper surface of the median nerve. One group will receive electrical stimulation and another won't. The investigators use electromyography, cross-section area of median nerve, visual analog scale, Boston Carpal Tunnel Syndrome Questionnaire, six-item scale, The disabilities of the arm, shoulder and hand score and Jamar grip dynamometer as outcome measurements. The results gathered from two experimental groups will be compared with the data from the control group whose participants only receiving local steroid injection once in the first week. The participants are all above 18 years old and complain of illness for a least 3 months without any surgery or local injection for a least 1 year. The investigators set up strict exclusive criteria and sample size estimation is 70.

ELIGIBILITY:
Inclusion Criteria:

1. All participants are must above 20 years old,
2. All participants are willing to join and can be cooperated with all the interviews and examinations.
3. The symptoms are compatible with carpal tunnel syndrome, including numbness, pain, paresthesia, tingling, burning sensation over a least 2 fingers and hand motor limitation which are dominated by median nerve.These symptoms have to sustain for more than 3 months and be diagnosed by electromyography, physical examination and physicians.
4. Those who underwent local injection including glucose, steroid or anaphylaxis will be recruited if the treatments finished more than a year.

Exclusion Criteria:

1. symptoms due to radiculopathy (When the patient also complains of symptoms radiating to the elbow or neck movement pain, the orthopedic doctor will make the definite diagnosis. )
2. Those who underwent decompression surgery.
3. CTS due to traumatic injury (confirmed by image)
4. Those who underwent local injection within a year.
5. CTS due to rheumatoid arthritis
6. CTS due to cancer
7. CTS due to peripheral artery occlusive disease
8. Those who have past history of psychosis.
9. Pregnancy(every woman will be confirmed by urine pregnancy test)

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2016-08; Primary Completion 2017-08 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
pain assessed on visual analog scale | 24 weeks
Boston Carpal Tunnel Syndrome Questionaire | 24 weeks
The 6-item CTS symptoms scale | 24 weeks
cross sectional area(CSA) of the median nerve | 24 weeks
  CSA of the median nerve below the distal wrist crease which is measured by the ultrasound(transverse view )
hand grip power | 24 weeks
  Jamar Hand grip Dynamometer as the measuring tool
The Disabilities of the Arm, Shoulder and Hand (DASH) Score | 24 weeks
compound muscle action potential(CMAP) | 24 weeks
  The CMAP is a summated voltage response from the individual muscle fibre action potentials and measured in millivolts (mV).
Wrist-palm sensory nerve conduction velocity(Wrist-palm SNCV) | 24 weeks
  Wrist-palm SNCV (m/s) = distance between stimulation site 1 and site 2 (mm)/[latency wrist- latency palm(ms)].
motor nerve conduction velocity(MNCV) | 24 weeks
  MNCV (m/s) = distance between stimulation site 1 and site 2 (mm)/[latency site 2 - latency site 1 (ms)].
sensory nerve action potential(SNAP) | 24 weeks
  The sensory nerve action potential (SNAP) is obtained by electrically stimulating sensory fibres and recording the nerve action potential at a point further along that nerve.

IPD SHARING:
Plan to Share IPD: No